CLINICAL TRIAL: NCT07317193
Title: DEFINING THE GENETIC DRIVERS OF ADULT-ONSET CHOLESTATIC LIVER DISEASE
Acronym: FIRST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Luisa Ronzoni, Principal Investigator, Medical Doctor, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FIRST
Record Dates: First submitted 2025-12-18; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cholestatic Liver Disease; Progressive Familial Intrahepatic Cholestasis
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of the Diagnostic Yield of WGS in Adult Patients with Idopathic Cholestasis (Experimental): The FIRST study is a single-center, non-pharmacological, interventional investigation that aims to determine the diagnostic yield of Whole Genome Sequencing (WGS) in adult patients with unexplained cholestatic liver disease or with atypical clinical presentations (such as particular forms of PSC or PBC). The study design involves enrolling 60 patients ("Cases") who undergo WGS on peripheral blood samples, a procedure considered extra standard of care.
  Interventions: Other: Advanced Whole Genome Sequencing to Identify Rare Pathogenic Variants in Unexplained Cholestatic Liver Disease

INTERVENTIONS:
Other: Advanced Whole Genome Sequencing to Identify Rare Pathogenic Variants in Unexplained Cholestatic Liver Disease — The intervention consists of advanced genetic analysis to identify the presence of rare harmful variants in genes known to be associated with cholestasis or in other genes related to liver disorders. The results from the cases will be compared with WGS data from a large group of 1025 healthy controls (previously collected within the FOGS study) to assess the enrichment of these variants. The primary objective is to establish the prevalence of pathogenic variants, while secondary objectives include identifying new potential genetic determinants to improve diagnostic accuracy and optimize the clinical management of these complex conditions.

SUMMARY:
Cholestatic disease in adults comprises a heterogeneous group of conditions characterized by intra- or extrahepatic alterations of bile flow that can lead to fibrosis or hepatic decompensation. Due to the heterogeneity of clinical manifestation, which is sometimes very subtle, diagnosis based on clinical, histological, and radiological evaluation is often very complicated. Genetic testing can be helpful in identifying the cause of the clinical phenotype, thereby allowing for targeted follow-up adequate to the patient's specific characteristics and risk factors. Although the utility of genetic analysis has been well documented for other liver diseases or in pediatric cohorts of children with cholestatic disease, the use and benefits of genetic testing in adults with cholestatic disease are still little explored and investigated. In this context, through the use of whole-genome sequencing (WGS), the FIRST project aims to evaluate the role of rare genetic variants in the pathogenesis of cholestatic disease and the utility of WGS in defining a genetic diagnosis.

ELIGIBILITY:
Inclusion Criteria:

Cases:

* Adults, aged > 18 years with:

  1. persistent or intermittent elevations in serum alkaline phosphatase (ALP) or gamma-glutamyltransferase (GGT) for at least six months not explained following standard diagnostic assessment adhering to the guidelines of the European Association for the Study of the Liver (EASL), or with a positive family history of unexplained cholestasis or hepato-biliary cancer, negative to previous genetic tests (targeted panel for PFIC genes or WES);
  2. primary sclerosing cholangitis (PSC) with unusual features: small-duct PSC, non-typical radiological findings according to radiological guidelines on PSC, absence of concomitant inflammatory bowel disease, negative to previous genetic tests (targeted panel for PFIC genes or WES) or who didn't perform previous genetic test;
  3. primary biliary cholangitis (PBC) without specific anti-mitochondrial antibodies, negative to previous genetic tests (targeted panel for PFIC genes or WES) or who didn't perform previous genetic test.
* Signature of informed consent

Controls:

-Blood donors (age 18-65 years) without clinical signs of liver diseases based on the collected clinical parameters: anthropometric (BMI>18 and <25), haematological (Hb, white blood cells, platelets within the reference range), biochemical traits (albumin, bilirubin, AST, ALT, GGT, ALP within the reference range), medical history (negative for chronic or concomitant diseases, including immunological diseases)

Exclusion Criteria:

Cases:

* Patients who do not possess the above inclusion criteria or have at least one of the following exclusion criteria:
* an already known genetic diagnosis explaining the clinical phenotype
* affected by other causes of liver disease such as viral or autoimmune hepatitis

Controls:

-Blood donors with clinical signs of liver diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint: Diagnostic Yield of Whole Genome Sequencing (WGS) in Adult Patients with Unexplained or Atypical Cholestasis | 9 months
  The Primary Endpoint is the determination of the prevalence of pathogenic variants in genes already known to be involved in genetic cholestasis, effectively assessing the diagnostic yield of the WGS approach in adult patients with unexplained or atypical cholestasis.

SECONDARY OUTCOMES:
Investigating New Genetic Determinants: Prevalence of Rare Variants in Liver-Related Genes | 9 months
  The Secondary Endpoint aims to establish the prevalence of rare harmful variants in a wider range of liver-related genes, such as those associated with mitochondrial hepatopathies, metabolic disorders, and ciliopathies. This aims to gain insights into pathogenesis and to identify new potential genetic determinants of the condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Istituto di Ricovero e Cura a Carattere Scientifico di natura pubblica, Milan, Milano, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT07317193/Prot_SAP_000.pdf